CLINICAL TRIAL: NCT04154397
Title: Enhancement of Posture Training Effectiveness With Error-enhancing Feedback and Cerebellar Stimulation
Brief Title: Posture Training and Cerebellar Stimulation in Elderly People
Acronym: P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MOST 105-2314-B-006 -014 -MY3
Record Dates: First submitted 2019-10-28; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Transcranial Electrical Stimulation
Keywords: Motor learning; Cerebellum transcranial electrical stimulation; Postural balance; Error feedback; Electroencephalography; Elderly

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- error-enhancing feedback (No Intervention): The project of the first arm was to investigate how visualized error size affects postural training effect of the elderly, with a particular focus on error amplification strategy to optimize training benefits for postural training that favors the use of feedback mechanism on postural control and error correction. All participants were randomly assigned into the control and error amplification groups. The control group was trained to remain static stance on the stabilometer with visual guidance that displayed the target signal and tilting angle of the stabilometer. For the error amplification group, they were trained with the same postural paradigm, except that the visual guidance was virtually manipulated so that the participants visually perceived twice of the execution errors during stabilometer stance. We contrasted training benefits between the two groups after completion of eight training trails of 1 minute.
- positive cerebellar transcranial stimulation (Experimental): The project of the second arm was to investigate the training benefits of using combined cerebellar transcranial direct current stimulation and visual error amplification on postural training during static stabilometer stance, in reference to sole visual error amplification. A particular focus was training-related alterations in error correction strategy and underlying cortical plasticity for postural balance.They were randomly assigned into the control (traditional error amplification)and cerebellar transcranial direct current stimulation groups. Both groups were trained to remain static stance on the stabilometer with visual guidance that displayed the target signal and tilting angle of the stabilometer. Under the condition of visual feedback without error amplification, we again contrasted training benefits between the two groups after completion of eight training trails of 1 minute.
  Interventions: Device: cerebellar transcranial stimulation
- sham cerebellar transcranial stimulation (Experimental): The project of the third arm was to investigate the training benefits of using combined cerebellar transcranial random current stimulation and visual error amplification on postural training during static stabilometer stance, in reference to sole visual error amplification. A particular focus was training-related alterations in error correction strategy and underlying cortical plasticity for postural balance. All participants were randomly assigned into the control (sham stimulation) and cerebellar transcranial random current stimulation and visual error amplification (ES) groups. Both groups were trained to remain static stance on the stabilometer with visual guidance that displayed the target signal and tilting angle of the stabilometer. Under the condition of visual feedback without error amplification, we again contrasted training benefits between the two groups after completion of eight training trails of 1 minute.
  Interventions: Device: cerebellar transcranial stimulation

INTERVENTIONS:
Device: cerebellar transcranial stimulation — Feedforward-based training benefits from a dynamic postural task by application of cerebellum transcranial electrical stimulation (ctDCS) of different modes (direct current vs. noise vs. sham) were administered using a one-channel direct current stimulator (NeuroConn DC-Stimulator PlusTM) with study mode enabled for single blinding. Following the baseline trial of posture tracking, participants of three groups were seated in a chair for 20 min to receive either active or sham cerebellar tDCS prior to the posture tracking and transfer test phases.
  Arms: positive cerebellar transcranial stimulation; sham cerebellar transcranial stimulation

SUMMARY:
Motor learning relies on both feedback and feedforward mechanisms to keep progressive optimization of motor behaviors in a coordinated manner. Error correction based on the fronto-parietal loop is subject to error information inherent within visual feedback. On the other hand, cerebellar activity for restoration of efferent copy involves in operation of feedforward mechanism. Therefore, the amount of error feedback and excitation of cerebellum are keyed to effectiveness of motor learning. Although postural training is of empirical value to prevent falling from the elderly, yet none of previous studies have ever been devoted to improve effectiveness of postural training via manipulations of visual error feedback and cerebellar stimulation.

From the aspect of cognition-motor interaction, the present proposal is a three-year project intended to promote effectiveness of postural training for the elderly. In the first year, feedback-based training benefits from a dynamic postural task under the conditions of different visual size of error feedback (error-reducing feedback, error-enhancing feedback, and fixed error feedback) will be contrasted. In the second year, feedforward-based training benefits from a dynamic postural task by application of cerebellum transcranial electrical stimulation (ctDCS) of different modes (direct current vs. noise vs. sham) will be contrasted. In the third year, the proposal will examine whether postural training with combined approach (error-enhancing feedback and ctDCS) could result in a superior training benefit to those of error-enhancing feedback alone and ctDCS alone approaches. In addition to innovative training intervention, this proposal will make use of current non-linear analyses on EEG signals and postural sway with graph analysis and heading analysis, respectively. It is expected to gain additional insight into behavior and brain mechanisms underlying learning-related changes with the postural training, potentially lending to a more effective training paradigm for postural stability of the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Age above 60 years old healthy older adults without a history of falls.
* Able to understand and give informed consent.
* The Mini-Mental State Examination test score above 25-30.
* Lower limb muscle strength is evaluated as G grade
* The corrected visual acuity was within the normal range.

Exclusion Criteria:

* Any known history of mental illness
* Any neuromuscular or degenerative neurological disease(ex:stroke、SCI、TBI...etc)
* Any known history of cerebral cerebellar disease or intracranial metal implants.
* Weak of hearing or wearing a hearing aid

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Graph theoretical analysis of EEG functional network | through study completion, an average of 1 year
  Graph theory will characterize EEG functional connectivity and brain network efficiency regarding to brain mechanisms for practice-related leaning transfer.This project introduced EEG pattern analysis into the posture research project. It is expected to find out the changes in brain network efficiency and functional structure caused by posture training. It is a tool for understanding the neural mechanism of this project.

SECONDARY OUTCOMES:
heading analysis of center of pressure | through study completion, an average of 1 year
  Trajectories of central of pressure will be analyzed with stabilogram diffusion analysis to reveal behavior mechanisms for practice-related variations in feedback and feedforward process for error corrections.

CONTACTS AND LOCATIONS:
Overall Officials: Hwang Ing-Shiou, Phd, Study Chair — NCKU, Institute of Allied Health Sciences